CLINICAL TRIAL: NCT03219853
Title: Investigating Flavour-nutrient Learning in Humans Using Selenium-enriched Parsnips
Brief Title: Investigating the Sensory Effects of Selenium-enriched Parsnips.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Collaborators: Fera Science (Unknown); Institute For Agri-food Research and Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NUHEALTH-AM01-SELENIUM
Record Dates: First submitted 2017-06-21; First posted 2017-07-18 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Food Sensory Perception; Selenium Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower selenium-status (Experimental)
  Interventions: Dietary Supplement: selenium enriched parsnips; Dietary Supplement: Conventional parsnips
- higher selenium (Experimental)
  Interventions: Dietary Supplement: selenium enriched parsnips; Dietary Supplement: Conventional parsnips

INTERVENTIONS:
Dietary Supplement: selenium enriched parsnips — Parsnips which have been grown in a selenium enriched environment
Dietary Supplement: Conventional parsnips — Parsnips which have been grown in a conventional environment

SUMMARY:
Study aims to investigate 2 topics:

1. Flavour-Nutrient Learning (FNL) FNL proposes that personal food preferences may be influenced by unconscious mechanisms which operate to ensure the safeguarding of individual nutrient levels. The theory postulates that food preferences may change over time to address changing nutritional status (Yeomans, 2012).

   This study aims to explore FNL in humans by investigating the preferences of participants with low and high blood-selenium levels in relation to selenium-enriched parsnips. Participants will be investigated in a two-week trial in which they will undertake two food sensory tests: one before, and one after, the two-week period where they will incorporate provided parsnips into their diet.

   Some provided parsnips will contain higher levels of selenium than others, neither the participants nor the lead researcher will know which type of parsnip each participant receives.

   It is hypothesised that the second food sensory test, performed after the intervention period, will show that participants of lower initial blood-selenium levels will demonstrate an increased liking for the selenium-enriched parsnips. This may demonstrate possible FNL in humans.
2. Relationship between selenium intake & plasma selenium-status. This study will also examine the relationship (if any) between the selenium intake of all participants via the different types of parsnips, and their individual blood-selenium levels.

This will be assessed via blood tests before, during and after the trial in order to observe the blood-selenium levels of each participant.

It is hypothesised that the blood-selenium levels of participants of lower initial selenium readings will be the most improved upon consumption of selenium-enriched parsnips.

DETAILED DESCRIPTION:
1. FNL Despite a wealth of animal studies (Amanoel et al, 2016; Bach et al, 2012), human FNL research is in relative infancy.

   This study intends to investigate FNL in humans by exploring preferences of participants of different selenium-status regarding selenium-enriched parsnips, with non-enriched parsnips and other root vegetables to be used as comparators.

   Participants will be assessed by means of food sensory tests and blood analysis before, during and after the trial period.

   The trial aims to recruit 26 lower selenium-status participants of initial selenium-status approx. 70μg/L, and 26 higher selenium-status participants of initial selenium-status approx. 100μg/L (n=52). (Initial screening sample approx. n=120.) On initial screening, potential participants recording a selenium-status of under 28μg/L or over 400μg/L will be excluded (and their GP informed) for safety reasons.

   Re parsnips:

   Selenium-enriched parsnips: Se content approx. 0.30ppm. Placebo comparator: non-selenium-enriched parsnips: Se content approx. 0.06ppm. Treatment portion: 200g fresh weight per day for 14 days. Comparator vegetables: potato, celeriac, turnip.
2. Relationship between selenium intake & plasma selenium-status. This study will also investigate the relationship, if any, between the selenium intake of all participants via the different types of parsnips and their individual selenium status. This will be assessed via blood tests before, during and after the trial in order to observe plasma-selenium status.

This is deemed an important area for research as research suggests a trend towards selenium deficiency in the United Kingdom population (SACN, 2013). It is hoped the current study may inform the debate regarding the potential of improving United Kingdom's population selenium status via selenium-fortified foods.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of either gender, aged over 18 years.
2. Willingness and ability to provide blood samples, consume parsnips daily for 2 weeks, and carry out 2 sensory tests, as described in the Participant Information Sheet.
3. Generally healthy, meaning that if health issues such as hypertension, diabetes, arthritis etc. are present, they are well controlled by appropriate treatments.

Exclusion Criteria:

1. Under 18 years.
2. Difficulties with chewing or swallowing.
3. Taste disorders.
4. Allergies to parsnips.
5. Impairments which may prevent mental understanding of trial, or informed consent from being given.
6. Taking supplements providing more than 60µg Se per day
7. Initial analysed selenium status of less than 28μg/L.
8. Initial analysed selenium status of over 400μg/L.
9. Any other condition that in the view of the participant's General Practitioner (GP) may make the participant unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-12-14 (Estimated); Study Completion 2017-12-14 (Estimated)

PRIMARY OUTCOMES:
Food sensory perception | Baseline & post 14 weeks supplementation
  change from baseline sensory perception of food samples

SECONDARY OUTCOMES:
Selenium status | Baseline, post 7 days supplementation ad post 14 days supplementation
  Change from baseline selenium status

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided